CLINICAL TRIAL: NCT06199037
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability and Pharmacodynamics of Intravenous Administration of SHR-1707 In Patients With Mild Cognitive Impairment Due to Alzheimer's Disease or Mild Alzheimer's Disease
Brief Title: Safety and Pharmacodynamics of SHR-1707 in Alzheimer's Disease Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1707-201
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-12

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: SHR-1707 compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1707 (Experimental)
  Interventions: Drug: SHR-1707
- SHR-1707 placebo (Placebo Comparator)
  Interventions: Drug: SHR-1707 placebo

INTERVENTIONS:
Drug: SHR-1707 — 1 cohort of Mild Cognitive Impairment Due to Alzheimer's Disease or Mild Alzheimer's Disease patients will receive SHR-1707 injection
  Arms: SHR-1707
Drug: SHR-1707 placebo — 1 cohort of Mild Cognitive Impairment Due to Alzheimer's Disease or Mild Alzheimer's Disease patients will receive SHR-1707 placebo injection
  Arms: SHR-1707 placebo

SUMMARY:
Evaluate the Safety, Tolerability and Pharmacodynamics of Intravenous Administration of SHR-1707 In Patients with Mild Cognitive Impairment Due to Alzheimer's Disease or Mild Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥50 and ≤85 on the date of signing the informed consent, males or females;
2. BMI≥18kg/m2 and ≤32 kg/m2, weight ≥45 kg且≤100 kg at screening or baseline；
3. must meet the diagnostic criteria for MCI due to AD or mild AD;
4. The total score of HAMD-17 should be ≤10 scores at screening;
5. The score of Hachinski ischemic scale should be ≤4 scores at screening;
6. amyloid PET scan results from the central laboratory confirmed the presence of pathological changes in AD;
7. Agreed to test ApoE genotype;
8. Have a stable caregiver; where symptomatic drugs for AD is used, they must be stable for at least 1 months prior to the screening visit;

Exclusion Criteria:

1. Cognitive impairment of subjects due to other medical or neurological factors (other than AD);
2. History of stroke or transient ischemic attack, seizures, or other unexplained loss of consciousness within the past year;
3. Any psychiatric diagnosis that may interfere with the subject's cognitive assessment;
4. Cannot tolerate MRI or has contraindications to MRI, has significant lesions shown on MRI during screening, or has other conditions that the investigator believes may bring a significant risk to the subject;
5. Patients who had severe trauma or had undergone surgery within 6 months prior to screening, or were scheduled to undergo surgery during the trial;
6. History of moderate (3b) or severe renal failure or insufficiency;
7. Uncontrolled hypertension: systolic blood pressure > 160mmHg and diastolic blood pressure >100mmHg during screening or baseline;
8. 12-lead ECG showed QTcF >450ms for male and >470ms for female during screening;
9. History of hypoglycemic coma or uncontrolled diabetes 6 months prior to the screening period;
10. Thyroid dysfunction；
11. Had unstable or clinically significant cardiovascular disease within 1 year prior to the screening period, had or currently has atrial fibrillation;
12. History of malignancy within 5 years prior to screening;
13. Patients with clinically significant systemic immunosuppression due to the persistent effects of immunosuppressive drugs;
14. Human immunodeficiency virus antibody (HIV-Ab), treponema pallidum antibody and hepatitis C virus antibody (HCV-Ab) were positive during screening.Hepatitis B active subjects [Hepatitis B virus surface antigen (HBsAg) positive with HBV DNA > upper limit of normal]
15. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeding 3 times ULN, or total bilirubin exceeding 2 times ULN
16. Folic acid or vitamin B12 below the lower limit of normal
17. coagulation disorders
18. According to the investigators, the subjects were suicidal or had committed suicidal behaviour in the six months before the screening period;
19. Severe visual or hearing impairment, unable to cooperate with the completion of the scale;
20. A woman who is pregnant, or a woman of childbearing potential whose pregnancy test results are positive, or who is breastfeeding; or has a plan to have a child, unwilling or unable to take effective contraceptive measures within 30 days prior to the screening period or six months after the last use of the investigational drug.
21. History of drug abuse or addiction;
22. Three months prior to the randomization period or planned to use dual antiplatelet or anticoagulant drugs during the trial;
23. Received any passive immunotherapy or other long-acting biologics used to prevent or delay cognitive decline within 3 months prior to screening;
24. Investigators and relevant staff of the research Centre or others directly involved in programme implementation;
25. The investigator considers that there are any circumstances that would cause the subject to be unable to complete the study or pose a significant risk to the subject or other factors that would interfere with the subject's ability to complete the study evaluation.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-06-24 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in intracerebral Aβ deposition at Week 26 as assessed by brain Aβ PET | Week 26

SECONDARY OUTCOMES:
To assess the number of patients with adverse events (AEs) | week 26
To assess the number of patients with clinically significant change from baseline in vital signs values | week 26
To assess the number of patients with clinically significant change in physical examination | week 26
To assess the number of patients with clinically significant change from baseline in laboratory examination | week 26
To assess the number of patients with clinically significant change from baseline in 12-ECG values | week 26
To assess the number of patients with clinically significant change in brain MRI | week 26
To assess the ADA | week 26
To assess the number of patients with adverse events (AEs) | week 52\week 78
To assess the number of patients with clinically significant change from baseline in vital signs values | week 52\week 78
To assess the number of patients with clinically significant change in physical examination | week 52\week 78
To assess the number of patients with clinically significant change from baseline in laboratory examination | week 52\week 78
To assess the number of patients with clinically significant change from baseline in 12-ECG values, | week 52\week 78
To assess the number of patients with clinically significant change in Head brain MRI | week 52\week 78

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated hospital of USTC, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided